CLINICAL TRIAL: NCT06463431
Title: A Trial for An Integrated Cognitive Behavioural Therapy to Treat PTSD and Sexually Transmitted Infections Among Gay, Bisexual, and Other Men Who Have Sex With Men
Brief Title: Cognitive Processing Therapy to Treat PTSD and Sexually Transmitted Infections Among Men Who Have Sex With Men
Acronym: CPT-T
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Toronto Metropolitan University (Other)
Responsible Party: Principal Investigator, Trevor Hart, Professor, Toronto Metropolitan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: REB 2024-251; 151412 (Other Grant/Funding Number: Toronto Metropolitan University); 152308 (Other Grant/Funding Number: CIHR)
Record Dates: First submitted 2024-03-18; First posted 2024-06-17 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Stress Disorders, Post-Traumatic; Sexually Transmitted Infection (STI) Prevention
Keywords: Cognitive Processing Therapy; men who have sex with men; gay bisexual queer men; gay men; post traumatic stress disorder; Cognitive Behavioral Therapy; sexually transmitted blood borne infections; sexual risk; prevention
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Sexually Transmitted Diseases; Homosexuality | interventions — 2-cyclohexylidenhydrazo-4-phenyl-thiazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cognitive Processing Therapy (Experimental): The intervention will consist of 14 90-minute weekly virtual sessions of CPT with a study therapist.
  Session 1: Discuss sexual history/goals regarding PTSD and STBBI risk reduction, including reducing CAS, using medications to treat HIV/bacterial STBBIs, & providing education about the benefits of using PrEP Session 2: Review the cognitive model for CPT and the index trauma Sessions 3-7: Address problematic appraisals of the index trauma, maladaptive thoughts, and the experience and expression of natural emotions. Teach cognitive intervention skills to facilitate cognitive & emotional change Sessions 8-12: Discuss/challenge beliefs regarding safety, trust, power/control, esteem, & intimacy Session 13: Identify how participant's changed beliefs may affect sexual decision making, CAS, and substance use in sexual situations Session 14: Discuss relapse prevention/goals for progress regarding PTSD, substance use, & STBBI risk reduction
  Interventions: Behavioral: Cognitive Processing Therapy

INTERVENTIONS:
Behavioral: Cognitive Processing Therapy — We propose a conceptual model for the relationship between PTSD, substance use, & sexual risk behaviour wherein using substances to avoid posttraumatic cognitions & affect leads to risky sexual behaviour through impaired safer sex negotiation. These mechanisms are consistent with the theory underlying CPT. Behaviourally, substance use (and potentially risky sexual behaviour) is negatively reinforced through avoiding unwanted negative affect. Cognitively, PTSD-based predictions may generate unrealistic risk appraisals that contribute to sexual risk. CPT addresses these specified pathways by a) identifying how trauma leads to maladaptive beliefs about the self, others, & the future, b) cognitive interventions to address these beliefs, & c) an overall trauma-focused orientation that addresses cognitive, affective & behavioural avoidance, using cognitive restructuring to lead to more realistic/adaptive beliefs, less cognitive/affective avoidance, & more goal-directed approach behaviours.
  Other Names: CPT

SUMMARY:
Gay, bisexual, queer, and other men who have sex with men (GBM) continue to bear a disproportionate burden of the sexually transmitted and blood-borne infections (STBBI), largely attributable to efficient transmission during condomless anal sex (CAS; Baggaley et al., 2010). In 2022, GBM accounted for 38.1% of new HIV diagnoses in Canada (Public Health Agency of Canada, 2023). Incidence of syphilis, chlamydia and gonorrhea have risen among men who have sex with men (MSM), especially among HIV+ GBM living in Canadian urban centres, including Toronto and Quebec (Public Health Agency of Canada, 2022). Post-traumatic stress disorder prevalence is also higher among GBM than among heterosexual men (Roberts et al., 2010). Post-traumatic stress disorder (PTSD) is a risk factor for CAS and related STBBI among GBM (O'Cleirigh, 2019). Despite the strong association between PTSD and STBBI risk among GBM, no studies have examined the efficacy of PTSD treatment on STBBI risk among GBM. PTSD may also increase substance use in sexual situations, another risk factor for STBBIs among GBQM (Semple et al., 2011; Elkington et al., 2010). Substance use tends to follow PTSD because alcohol and other substances are often used to self-medicate trauma symptoms (as an avoidant coping strategy) in interpersonal situations (Tan et al., 2021). Alcohol and substance use in sexual situations are consistent risk factors for CAS among Canadian GBQM (Lambert et al., 2011), and are associated with higher HIV incidence. Due to consistent data linking substance use to STBBI risk, it has been suggested that incorporating alcohol and substance use treatment into sexual risk reduction counselling (Koblin et al., 2006; Parsons et al., 2005; Shoptaw & Frosch, 2000) may increase the efficacy of STBBI prevention efforts for GBQM. PTSD is highly treatable via cognitive-behavioural therapies, including by Cognitive Processing Therapy (CPT; Benight & Bandura, 2004; Monson & Shnaider, 2014; Watkins et al., 2018).

The present study will provide preliminary feasibility and acceptability data for a novel and innovative STI/HIV prevention intervention for GBQM. This intervention builds upon empirically supported treatments for PTSD, including PTSD-related substance use, by adding risk reduction counselling to reduce sexually transmitted infections (STI) and HIV sexual risk behaviour. The present study will provide trial data for a novel and innovative STBBI prevention psychotherapy for GBM that could be administered by mental health providers across Canada. The intervention will consist of 14 90-minute sessions of an integrated cognitive-behavioural approach using CPT to treat PTSD and to reduce STBBI risks among GBQM. The primary outcome will be condomless anal sex with casual partners. The secondary outcomes will be PTSD prevalence, trauma symptoms, problematic substance use, sexual risk, and PTSD-related avoidance of negative thoughts and feelings.

This psychotherapy intervention will build upon empirically supported interventions to reduce HIV risk.

ELIGIBILITY:
Inclusion Criteria:

* Live in Ontario or Quebec (able to travel to Toronto Metropolitan University or CLSC de Cote-des-Neiges, respectively)
* Identify as a man
* Are over 18 years of age
* Have had anal sex without a condom with a person assigned male at birth in the past 3 months
* Have experienced symptoms consistent with a diagnosis of PTSD
* Are able to read, speak, and understand English

Exclusion Criteria:

* if a 14-session protocol is deemed inappropriate for their treatment needs (e.g., psychotic or bipolar disorders not well-managed by medications)
* if either our assessors or therapists identify that a participant's ability to respond to study measures is compromised by mental or physical disabilities or inability to speak and understand English

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants must report self-identifying as a man (cisgender or transgender)
Enrollment: 56 (Estimated)
Dates: Start 2025-03-31 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Condomless anal sex (CAS) with casual partners, based on response at 6 months. | 3-months following final treatment session
  Participants will indicate frequency of CAS and number of casual sex partners, defined as partners of less than a 6-month duration for 1) insertive and receptive anal sex and vaginal or frontal sex both with and without a condom, in the past 3 months.

SECONDARY OUTCOMES:
PTSD Measures | baseline, post-intervention (an average of 16-18 weeks after baseline), 3-month follow-up
  PTSD Scale-5 (CAPS-5). The CAPS-5 will be our primary measure of PTSD. The CAPS-5 includes a lifetime trauma checklist and questions about stressor exposure, which will be used to ensure that participants meet the DSM-5 criterion of traumatic stressor criteria exposure that is required for diagnosis. The CAPS-5 yields a continuous measure of PTSD severity, as well as diagnostic status. The psychometric properties of the CAPS-5 have been well-established.
Self-Report Measures - PTSD | baseline, post-intervention (an average of 16-18 weeks after baseline), 3-month follow-up
  PTSD. The Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5) is a well-validated measure of PTSD severity. The Impact of Events - Revised scale will also be used to evaluate our mediator of avoidance of negative cognitions and affect and provide additional data on participants' trauma.
Self-Report Measures - Sexual behavior | baseline, post-intervention (an average of 16-18 weeks after baseline), 3-month follow-up
  Self-report: Frequency and number of sexual partners
Change in Clinical diagnosis and Severity of Mental Health Symptoms | baseline, post-intervention (an average of 16-18 weeks after baseline), 3-month follow-up
  The Structured Clinical Interview for DSM-5 Disorders (SCID-5) will be used to determine whether participants meet diagnostic criteria for PTSD disorder or any other psychological disorder. A subset of 20% of randomly selected baseline assessments will be reviewed by a second diagnostician for reliability.
Cumulative incidence of bacterial STIs and incidence of HIV and viral hepatitis | baseline, post-intervention (an average of 16-18 weeks after baseline), 3-month follow-up
  Laboratory specimens will be collected via blood tests, and throat and rectal swabs. We will also ask for self-report of HIV/STI incidence in the last 6 months.
Self-Report Measures - Substance Use. | baseline, post-intervention (an average of 16-18 weeks after baseline), 3-month follow-up
  To assess substance use and dependence problems, we will use the well validated and highly reliable World Health Organization Alcohol, Smoking and Substance Involvement Screening Test (WHO-ASSIST).
Qualitative Exit Interview | post-intervention (an average of 16-18 weeks after baseline)
  This is a structured interview that guides the participant through primary open-ended questions concerning their experience of the intervention. These questions are designed to solicit information of the acceptability of the intervention and the participant's satisfaction with intervention. A sample question is "Do you have any concerns about the program or recommendations for improvement?" The interview takes approximately 30 minutes to complete.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Toronto Metropolitan University, Toronto, Ontario
  - McGill University, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shoptaw S, Frosch D. Substance abuse treatment as HIV prevention for men who have sex with men. AIDS Behav. 2000;4(2):193-203.
- [Background] Parsons JT, Kutnick AH, Halkitis PN, Punzalan JC, Carbonari JP. Sexual risk behaviors and substance use among alcohol abusing HIV-positive men who have sex with men. J Psychoactive Drugs. 2005 Mar;37(1):27-36. doi: 10.1080/02791072.2005.10399746. PMID 15916249
- [Background] Koblin BA, Husnik MJ, Colfax G, Huang Y, Madison M, Mayer K, Barresi PJ, Coates TJ, Chesney MA, Buchbinder S. Risk factors for HIV infection among men who have sex with men. AIDS. 2006 Mar 21;20(5):731-9. doi: 10.1097/01.aids.0000216374.61442.55. PMID 16514304
- [Background] Lambert G, Cox J, Hottes TS, Tremblay C, Frigault LR, Alary M, Otis J, Remis RS; M-Track Study Group. Correlates of unprotected anal sex at last sexual episode: analysis from a surveillance study of men who have sex with men in Montreal. AIDS Behav. 2011 Apr;15(3):584-95. doi: 10.1007/s10461-009-9605-3. PMID 20033763
- [Background] Tan RKJ, Phua K, Tan A, Gan DCJ, Ho LPP, Ong EJ, See MY. Exploring the role of trauma in underpinning sexualised drug use ('chemsex') among gay, bisexual and other men who have sex with men in Singapore. Int J Drug Policy. 2021 Nov;97:103333. doi: 10.1016/j.drugpo.2021.103333. Epub 2021 Jun 24. PMID 34175526
- [Background] Elkington KS, Bauermeister JA, Zimmerman MA. Psychological distress, substance use, and HIV/STI risk behaviors among youth. J Youth Adolesc. 2010 May;39(5):514-27. doi: 10.1007/s10964-010-9524-7. Epub 2010 Mar 14. PMID 20229264
- [Background] Semple SJ, Strathdee SA, Zians J, McQuaid JR, Patterson TL. Drug assertiveness and sexual risk-taking behavior in a sample of HIV-positive, methamphetamine-using men who have sex with men. J Subst Abuse Treat. 2011 Oct;41(3):265-72. doi: 10.1016/j.jsat.2011.03.006. Epub 2011 May 8. PMID 21550758
- [Background] Benight CC, Bandura A. Social cognitive theory of posttraumatic recovery: the role of perceived self-efficacy. Behav Res Ther. 2004 Oct;42(10):1129-48. doi: 10.1016/j.brat.2003.08.008. PMID 15350854
- [Background] Roberts AL, Austin SB, Corliss HL, Vandermorris AK, Koenen KC. Pervasive trauma exposure among US sexual orientation minority adults and risk of posttraumatic stress disorder. Am J Public Health. 2010 Dec;100(12):2433-41. doi: 10.2105/AJPH.2009.168971. Epub 2010 Apr 15. PMID 20395586
- [Background] O'Cleirigh C, Safren SA, Taylor SW, Goshe BM, Bedoya CA, Marquez SM, Boroughs MS, Shipherd JC. Cognitive Behavioral Therapy for Trauma and Self-Care (CBT-TSC) in Men Who have Sex with Men with a History of Childhood Sexual Abuse: A Randomized Controlled Trial. AIDS Behav. 2019 Sep;23(9):2421-2431. doi: 10.1007/s10461-019-02482-z. PMID 30993478
- [Background] Baggaley RF, White RG, Boily MC. Infectiousness of HIV-infected homosexual men in the era of highly active antiretroviral therapy. AIDS. 2010 Sep 24;24(15):2418-20. doi: 10.1097/QAD.0b013e32833dbdfd. No abstract available. PMID 20827059
- See also: Study Webpage — https://hivprevlab.ca/research/resilience-and-sexual-health-empowerment-rise/